CLINICAL TRIAL: NCT04621162
Title: Evaluation of the Influence of Cognitive Variables in Hypoalgesia Generated by Motor Imagery: A Randomized Controlled Trial
Brief Title: Effects of Expectations on Hypoalgesia Produced by Mental Practice
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Autonoma de Madrid (Other)
Collaborators: Centro Universitario La Salle (Other)
Responsible Party: Principal Investigator, Roy La Touche Arbizu, Principal Investigator, Universidad Autonoma de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: uammadrid100
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Cognitive Change
Keywords: Motor imagery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Positive Expectations (initial) (Experimental)
  Interventions: Behavioral: Positive Expectations (initial)
- Negative Expectations (initial) (Experimental)
  Interventions: Behavioral: Negative Expectations (initial)
- Neutral Expectations (initial) (Placebo Comparator)
  Interventions: Behavioral: Neutral Expectations (initial)
- Positive Expectations (during intervention) (Experimental)
  Interventions: Behavioral: Positive Expectations (during intervention)
- Negative Expectations (during intervention) (Experimental)
  Interventions: Behavioral: Experimental: Negative Expectations (during intervention)
- Neutral Expectations (during intervention) (Placebo Comparator)
  Interventions: Behavioral: Neutral Expectations (during intervention)

INTERVENTIONS:
Behavioral: Positive Expectations (initial) — A positive expectation of the effect of motor imagery will be given before beginning the mental practice of imagination. "This task will generate hypoalgesia"
  Arms: Positive Expectations (initial)
Behavioral: Negative Expectations (initial) — A negative expectation of the effect of motor imagery will be given before beginning the mental practice of imagination. "This task will not generate hypoalgesia"
  Arms: Negative Expectations (initial)
Behavioral: Neutral Expectations (initial) — This group will act as a control. No expectations will be given that will influence the participant.
  Arms: Neutral Expectations (initial)
Behavioral: Positive Expectations (during intervention) — A positive expectation will be given during the performance of the mental practice. "This is working very well"
  Arms: Positive Expectations (during intervention)
Behavioral: Experimental: Negative Expectations (during intervention) — A negative expectation will be given during the performance of the mental practice. "This is working very bad"
  Arms: Negative Expectations (during intervention)
Behavioral: Neutral Expectations (during intervention) — This group will act as a control. No expectations will be given that will influence the participant.
  Arms: Neutral Expectations (during intervention)

SUMMARY:
The main objective of this research work is to evaluate and quantify the hypoalgesia generated by motor imagery influenced by the presence of expectations.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60
* Healthy and with no pain subjects

Exclusion Criteria:

* Any cognitive impairment that hindered viewing of audiovisual material.
* Difficulty understanding or communicating.
* Presence of systemic pathology, Central Nervous System or rheumatic disease.
* Inadequate understanding of the Spanish language to follow instructions for measuring and treatment.
* Collaboration of pregnant women.
* Underage subjects
* Subjects with pain at the time of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-12-30 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Pain pressure threshold | Change from baseline and immediately post-intervention
  Pressure Pain Threshold (PPT) is one of these tests and it is defined as the minimum force applied which induces pain. The measurement shall be carried out by using an algometer (pressure device that induces mechanical stimuli) is to standardize the amount of pressure applied in the neck region. The reliability of pressure pain thresholds according to raters or measurement frequencies is relatively high.
Thermal threshold | Change from baseline and immediately post-intervention
  This variable will evaluate three aspects. Cold detection threshold, heat detection threshold and heat pain threshold. A specialized and validated instrument is used which consists of a sensor with a resistance that raises and lowers the temperature in a controlled way between 20 and 50ºC.
Heart Rate | Change from baseline and immediately post-intervention
  Heart Rate will be measured by three electrodes located in the left area of the chest. One of the electrodes is placed in the middle zone while a second electrode is positioned on the lateral side, and a third one on the lower left side, below the first electrode.

CONTACTS AND LOCATIONS:
Locations (1):
- CSEU La Salle, Madrid, Spain